CLINICAL TRIAL: NCT02550327
Title: A Pilot Study of Gemcitabine, Nab-Paclitaxel, Cisplatin and Anakinra Treatment on Patients With Resectable or Potentially Resectable Pancreatic Adenocarcinoma (PDAC)
Brief Title: Gemcitabine, Nab-Paclitaxel, Cisplatin and Anakinra Treatment on Patients With Pancreatic Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 015-198
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: resectable; potentially resectable; Pancreatic adenocarcinoma; PDAC
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Cisplatin; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Experimental): All patients will receive Nab-paclitaxel, Gemcitabine, Cisplatin, and Anakinra given on Day 1 and 8 of a 21 day cycle (two weeks on with one week rest). Anakinra will be self-administered subcutaneously corresponding with chemotherapy.
  The patient will complete a total of 6 cycles of chemotherapy.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Cisplatin; Drug: Anakinra

INTERVENTIONS:
Drug: Nab-paclitaxel — 125 mg/m2
  Other Names: Abraxane
Drug: Gemcitabine — 1000 mg/m2
  Other Names: Gemzar ®
Drug: Cisplatin — 25 mg/m2
  Other Names: Platinol
Drug: Anakinra — 100 mg
  Other Names: Kineret

SUMMARY:
The objective of this study is to improve survival by the addition of anakinra to the chemotherapy combination of nab-paclitaxel, gemcitabine, and cisplatin in patients with resectable or potentially resectable pancreatic adenocarcinoma (PDAC). The primary endpoint of the study is to determine whether the combination of abraxane, gemcitabine, cisplatin, and anakinra will improve disease-free survival (DFS) and to determine the number of patients who meet or surpass 11.5 months of DFS.

The secondary objectives of this study are to evaluate the effect of anakinra when combined with the three-drug regimen of nab-paclitaxel, gemcitabine, and cisplatin on response rate and overall survival after diagnosis and adverse events of patients with resectable or potentially resectable PDAC. The investigators will use the benchmark of 24 months overall survival (OS) to determine how many patients meet or exceed this goal. The investigators will monitor, by survey, patients' health related quality of life while on treatment to determine if the addition of anakinra improves this measure.

DETAILED DESCRIPTION:
This is a single-arm, open-label pilot study. Patients will receive Nab-paclitaxel, gemcitabine, cisplatin and anakinra.

ELIGIBILITY:
Inclusion Criteria: A patient will be eligible for inclusion in this study if he or she meets all of the following criteria:

1. Male or female ≥ 18 years of age.
2. Suspected PDAC prior to diagnosis or histological diagnosis of adenocarcinoma of the pancreas confirmed by pathology. Mixed subtypes of adenocarcinoma are acceptable as long as majority of cells are ductal adenocarcinoma. Subjects with suspected PDAC are those without a biopsy and a pancreas mass which appears to be metastatic disease. These subjects will be enrolled prior to biopsy and then excluded if a diagnosis of pancreas cancer is not confirmed by histology.
3. American Joint Committee on Cancer (AJCC) Stage I-III Pancreatic carcinoma.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
5. Serum albumin ≥2.0 gm/dL.
6. Expected survival ≥6 months.
7. Adequate hematologic function as defined by:

   * Absolute neutrophil count (ANC) >1500/mm3
   * Platelets ≥70,000/mm3
   * Hemoglobin >9 g/dL (in the absence of red blood transfusion).
8. Adequate liver function, as defined by:

   * Serum total bilirubin ≤2 x ULN mg/dL, prior to initiation of treatment.
   * Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN).
9. Adequate renal function, as defined by serum creatinine ≤ 1.5 x ULN, or creatinine clearance ≥50 mL/min
10. All females of child bearing potential must agree to use contraception to avoid pregnancy throughout the study and for one month after the last dose.
11. Patients must be accessible for treatment and follow-up.
12. Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate. Patients may not be consented by a medical power of attorney.

Exclusion Criteria: A patient will be ineligible for inclusion in this study if he or she meets any of the following criteria:

1. < 18 years of age.
2. History of organ transplant.
3. Other malignancy within five years, unless the probability of recurrence of the prior malignancy is <5% as determined by the Principal Investigator based on available information.
4. Current, active immunosuppressive therapy such as cyclosporine, tacrolimus
5. Significant or uncontrolled congestive heart failure (CHF), myocardial infarction or significant ventricular arrhythmias within the last 6 months.
6. Active infection or antibiotics within 48 hours prior to study enrollment, including unexplained fever (temp > 38°C).
7. Other severe and/or uncontrolled medical conditions or other conditions that in the opinion of the investigator could affect the participation of the patient on the study.
8. Study consent form not signed.
9. Pregnant or nursing women.
10. Known HIV positive status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 2 Years
  determine the number of patients who meet or surpass 11.5 months of disease free survival

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  The use of a benchmark of 24 months overall survival will be used to determine how many patients meet or exceed this goal.
Quality of Life | 2 years
  The use of surveys will capture the patients' health-related quality life while on treatment to determine if the addition of anakinra improves this measure.
Toxicities and Adverse Events will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. | 2 years
  Toxicities and adverse events will be recorded from the of informed consent to 30 days following the last study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Becerra, MD, Principal Investigator — Baylor Research Institute/Texas Oncology
Locations (1):
- Baylor Charles A. Sammons Cancer Center, Dallas, Texas, United States